CLINICAL TRIAL: NCT02228876
Title: A Family Study of Copy Number Variations in Patients With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201403019RINA
Record Dates: First submitted 2014-08-18; First posted 2014-08-29 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This 3-year proposal is a family-based cohort study to establish a representative sample of probands with ASD and their parents with well-characterized environmental, clinical phenotypes, endophenotypes, and genetic data to conduct CNV experiments and the genotype-phenotype correlations. Based on our previous findings, probands with CNVs larger than 500kb has been identified and their families will be newly recruit in the present project to reveal the origin of the CNVs and reveal the clinical feature of the families. The significant findings in specific genes will conduct pathway analysis to reveal the etiology in ASD, providing further understanding in the disease.

DETAILED DESCRIPTION:
Due to its high prevalence, long-term impairment, high genetic component (heritability > 90%), and lack of effective prevention and treatment, ASD has been prioritized for genetic studies. However, despite extensive genetic research, there has been no any conclusive result mainly due to the clinical and genetic heterogeneity of ASD. Given the progress of CNV study in ASD, several challenges remain to be faced with, such as differences in phenotypic definition across different studies; a lack of population norms for CNVs, and a lack of consensus in methods for CNV detection and analysis. In the present study, the large segments of CNV found in ASD probands will be compared with standardized controls from National Center for Genome Medicine (NCGM), Academia Sinica to identify the possible CNVs. The other important issue of CNV research in ASD is to investigate whether the origin of CNVs are inherited or de novo. By collecting the complete background and revealing the CNVs of the parents and siblings, the origin of the CNVs will be uncovered in the present project. The candidate genes from important CNVs will be identified by pathway analysis. Gene expression will be conducted to confirm the pathogenic genes. Notably the present study will help bridge the gap to translate the bench findings to bedside to help early detection of ASD and pave the way developing effective treatment for ASD in the future.

Specific Aims:

With the above-mentioned rationale of this project and limited research budget from NSC, the ultimate goal of this project is to identify the important CNVs to reveal the pathogenic genes for ASD for future translational research in ASD and to prospectively characterize clinical features of ASD individuals with CNV.

The specific aims of this study are as follows,

1. To identify important and pathogenic CNVs by comparing the CNVs and CNPs of the controls provided by NCGM , Academia Sinica;
2. To assess parents and siblings of ASD patients who were found to have ~500 kb CNVs in our previous study using clinical, psychopathological, and social measures for family study and also to conduct CNV analysis in the families to determine the origin of the CNVs;
3. To conduct a follow-up assessments of clinical features, and social and neuropsychological functions of ASD probands with CNV to examine the phenotype changes over time;
4. To study the clinical phenotypes between de novo and inherited groups to reveal the pathogenic CNVs;
5. To conduct pathway analysis of genes involved in the CNVs, and to confirm the pathogenic genes by conducting gene expression analysis;
6. To investigate the associations of clinical phenotypes such as autistic tendency, and social impairments between (1) probands with/without CNVs/controls, and (2) probands/unaffected siblings/controls.

ELIGIBILITY:
Inclusion Criteria:

1. subjects have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV and ICD-10 criteria and ASD defined by the DSM-5, which was made by board-certificated child psychiatrists at the first visit and following visits;
2. their ages range from 3 to 30;
3. subjects have at least one biological parent;
4. both parents are Han Chinese; and
5. subjects and their biological parents consent to participate in this study for complete phenotype assessments and blood withdraw for genetic study.

Exclusion Criteria:

* if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, or Organic Psychosis.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on our preliminary CNV results of 339 probands, approximately 120 probands had been identified to have CNVs larger than 500kb. In the present project, the parents and siblings of the probands with CNVs larger than 500kb will be recruited (estimated sample size, parents = 200, siblings = 40) and reassess the ~120 probands.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of autism | 1 day
  Using the Autism Diagnostic Interview-Revised (ADI-R) to assess the developmental and behavioral aspects of autism, including reciprocal social interaction, communication, and repetitive behaviors and stereotyped patterns

SECONDARY OUTCOMES:
Diagnosis of psychiatric disorders | 1 day
  Using the Schedule for Affective Disorders & Schizophrenia (K-SADS-E) to assess the DSM-IV diagnosis of ADHD and other psychiatric disorders

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan